CLINICAL TRIAL: NCT03264924
Title: A Single-Centre, Feasibility Study to Promote Physical Activity Uptake and Adherence in Cardiac and Pulmonary Rehabilitation
Brief Title: Improving Physical Activity in Rehabilitation
Acronym: IPAiR
Status: Completed | Type: Observational
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Edge Hill University (Other)
Responsible Party: Sponsor
Other Study IDs: LiverpoolHeartNHS
Record Dates: First submitted 2017-06-16; First posted 2017-08-29 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Diseases; Pulmonary Disease; Chronic Obstructive Pulmonary Disease
Keywords: physical activity; motivation; behaviour change
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase A, Study One: Semi-structured interviews to investigate staff and patients' experiences of participating and facilitating cardiac and pulmonary rehabilitation.
- Phase A, Study Two: Focus group with rehabilitation stakeholders to discuss perceived feasibility and acceptability of the intervention design.
- Phase A, Study Three: Pilot of the intervention, using a group of exercise physiologists external to the community rehabilitation services.
  Interventions: Behavioral: IPAIR
- Phase B: Community rehabilitation service staff will participate in the intervention. Patients will then participate in the rehabilitaiton programme. Physical activity levels of patients will be recorded throughout the rehabilitation programme and for six months post-discharge. Qualitative and quantitative follow-up sessions will patients will take place at discharge (8 weeks after start of rehabilitation), and three and six months post-discharge.
  Interventions: Behavioral: IPAIR

INTERVENTIONS:
Behavioral: IPAIR — Motivational interview training
  Other Names: Motivational interview training
  Groups: Phase A, Study Three; Phase B

SUMMARY:
Cardiac rehabilitation is a programme of exercise and health advice for people recovering from heart disease. Pulmonary rehabilitation is a similar programme for people with chronic lung disease. For both groups of patients, taking part in rehabilitation can lead to improvements in health and well-being. However, only 30% of patients complete their agreed rehabilitation programme. This costs the NHS millions of pounds every year. This project aims to investigate whether a motivational-based intervention, underpinned by self-determination theory and motivational interviewing, will enable staff to encourage more patients to take part in physical activity (PA). Staff will be trained with the new communication skills and will then deliver the rehabilitation programme. The session content will not change, just the way in which staff speak to patients.

This will be a two-phase study. Phase A will take a qualitative approach collect patient and staff feedback about the current rehabilitation programme, before using this information to develop and pilot the intervention. Phase B will then assess the feasibility of the intervention within cardiac and pulmonary rehabilitation. Participants agreeing to take part in the phase B will be required to complete an interview and questionnaire at three time points. Patients' personal opinions of the programmes will be extremely important in discovering what can be done to improve rehabilitation for future participants.

The main objectives will be to look at whether the intervention increases the number of patients taking part in physical activity. The investigators plan to establish how much physical activity patients take part in whilst they are in rehabilitation, as well as once they have left the programme. This is why participants will be interviewed three and six months after they have finished their rehabilitation programme.

DETAILED DESCRIPTION:
Background and Rationale

Description of research questions and justification for undertaking the trial Cardiac Rehabilitation (CR) is an effective treatment for CHD and CVD patients, boasting a range of physiological and psychological benefits as well as lowering mortality and risk of secondary cardiac incidents. Despite the aforementioned benefits of CR attendance, uptake and adherence to CR remain inadequate, with cross-cultural surveys demonstrating that only 10-30% of eligible CR patients engage in such programmes. These poor levels of CR participation have been previously attributed to low referral rates amongst healthcare providers, however even within the 30% of eligible patients who become CR participants, the attrition rate is currently 50% and only 20% of attendees report long-term behavioural change. The lack of subsequent engagement with the desired adaptive behaviours is at a great cost to the National Health Service (NHS), with the cost of delivering a "good quality CR service" at £477 per patient and the average cardiac readmission costing £3637. Although physical activity (PA) has been demonstrated to reduce the risk of secondary cardiac incidents, 80% of CR patients fail to maintain regular habitual PA within the first year following a course of CR..

Similarly, Pulmonary Rehabilitation (PR) has been demonstrated to be an effective non-pharmacological intervention for COPD patients, and aims to return the patient to independent functioning, reduce disability and improve quality of life. The clinical conditions for which PR is routinely offered result in progressive loss of function over time. Therefore, any initial beneficial effects of a PR programme are likely to diminish over the subsequent eighteen months. Within this time period however, patients who complete PR have significantly greater quality of life, PA capacity, and fewer days in hospital relative to participants who do not participate in PR . Despite these benefits, uptake and adherence to PR is extremely problematic, with studies demonstrating that less than 50% of patients referred to PR will complete the course. Additionally, adherence rates reported in randomised controlled trials tend to be higher, so even this bleak estimate of adherence may be inflated.

Background Information

A commonality between CR and PR is the patients' participation in physical activity. Regular participation in physical activity (PA) reduces all-cause mortality by 30%, and can help to manage over 20 chronic conditions, including CHD, stroke, type 2 diabetes, cancer, obesity, mental health problems and musculoskeletal conditions. COPD patients' engagement in low-to-moderate intensity daily PA has been shown to enhance their cardiorespiratory health and ability for exertion, and reduce dyspnoea symptoms . Additionally, PA reduces cardiac mortality by 31%, and has been demonstrated to lower blood pressure, and increase 'good' cholesterol in cardiac patients. These effects occur through engagement in relatively low levels of activity: 30 minutes, five times per week.

Despite these far-reaching benefits, patients are less likely than non-symptomatic individuals to engage with PA. In 2015, a report by the Academy of Medical Royal Colleges portrayed PA as a 'miracle cure', which despite having a better disease risk reduction than many drugs, is often overlooked by healthcare providers and their patients. Worryingly, with the number of older people with multiple medical problems increasing rapidly, less than a third of UK adults over the age of 65 meet the minimum levels of PA.

Theoretical Underpinning

Motivation is a key component of behaviour change. With the focus on the motivational aspects of behaviour change in mind, Self-Determination Theory (SDT) has become an increasingly commonly used theory to design health behaviour change interventions . According to SDT individuals adopt or change behaviour on the basis of internal satisfaction and fulfilment, termed as intrinsic motivation. Alternatively, individuals are less likely to adopt or change behaviour when a reward or inducement provided by an external person is used to compel a person to act, known as extrinsic motivation. Environments that support intrinsic motivation optimise behavioural effort, persistence and performance. In contrast, environments that coerce through rewards serve to diminish behavioural effort, persistence and performance .

Previous SDT research has demonstrated that intrinsic motivation towards treatment is positively associated with adherence to medical regimes among people with chronic illnesses, attendance/involvement in an addiction treatment program, and long-term maintenance of weight loss among morbidly obese patients. Within physical activity research, intrinsic motivation has been found to be strongly associated with physical activity engagement. Similarly, increases in intrinsic motivation from pre- to post- exercise referral scheme significantly predicted greater adherence to the scheme as well as greater sports-related physical activity. The dense body of SDT research in health, including physical activity, suggests that interventions underpinned by SDT, should develop and support intrinsic motivation in order to optimally motivate engagement with PA.

Motivational interviewing (MI) is a method of strengthening personal motivation for change, and has been shown to be a promising approach for promoting health behaviour change in a number of contexts including physical activity promotion. MI comprises several techniques used by practitioners to facilitate behaviour change in patients. Some techniques focus on the content of the intervention, whereas others focus on techniques reflect the practitioner's interpersonal style of delivery. One of the primary roles the MI approach is to evoke the patient's arguments for change and to reduce their own arguments for not changing.

Research Critique

Motivational theories that inform behaviour change (for example, SDT) do not typically feed through to into instructor training programmes, particularly in clinical rehabilitation settings. Therefore, a significant limitation of motivational theory to date is its ability to be translated into clinical practice. Accordingly, it is important that attempts are made to ensure motivational theory is translated effectively in clinical practice in order to increase patients' motivation for physical activity uptake and adherence in cardiac and pulmonary rehabilitation. The current research, therefore, will combine a well-established motivational theory (i.e., Self-Determination Theory) with established motivational practice (i.e., Motivational Interviewing) in an attempt to integrate theory and practice, offsetting Ntoumanis et al's. claims that contemporary motivation research does not typically feed through to instructor programmes.

Previous researches aiming to increase physical activity motivation in rehabilitation have predominantly focused on interventions at an individual-level. Whilst it is important not to completely disregard this approach, the NHS rehabilitation setting is typically a place where clinicians have to facilitate sessions on a group-level. Furthermore, the NHS may not have the resources to provide the sufficient level of treatment fidelity that one-to-one approaches require in order to be successful. Therefore, the current research will equip clinicians with skills to be effective for increasing group-level physical activity motivation, as well as on an individual level.

Motivational-based intervention research for changing increasing physical activity behaviour in clinical rehabilitation settings has predominantly focused on intervention effectiveness for changing behavioural outcomes. However, the intervention development, delivery and content are not often reported, therefore, limiting the applied utility and replication of the intervention itself. As such, the current research will pilot and feasibly investigate the development of a motivational-based intervention. Doing so will provide a more nuanced understanding for motivating cardiac and pulmonary patients' uptake and adherence to physical rehabilitation activity. Such information would also be crucial for informing a future RCT trial.

ELIGIBILITY:
1. Inclusion criteria - Patients will be included when they enrol into cardiac and pulmonary rehabilitation programme due to heart disease or chronic obstructive pulmonary disease.
2. Exclusion criteria - They will be excluded if they have previously completed a cardiac/pulmonary rehabilitation programme.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac and pulmonary rehabilitation patients and staff.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage enrolment and attendance to rehabilitation | June 2018-February 2019.
  Measure of percentage enrolment and attendance to rehabilitation.

SECONDARY OUTCOMES:
Qualitative Impact Evaluation | June 2018-February 2019. Interviews will be conducted upon discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge
  Semi-Structured interview with patients and staff.
Treatment Self Regulation Questionnaire (Exercise) | June 2018-February 2019.Questionnaires will be completed upon admission to rehabilitation, discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge.
  The treatment self-regulation questionnaire (TSRQ) assessed autonomous and controlled reasons for participation in the program. The TSRQ has 18 item stems such as: "I am staying in the program because…", followed by several reasons that vary in the extent to which they represent autonomous regulation. An example of more controlled reasons are:"I feel like a failure if I don't". An example of more autonomous reasons are "I believe it's the best way to help myself." Each reason was rated on a 7-point scale ranging from not true at all to very true. Typically, the responses on the autonomous items are summed to form the autonomous regulation score (range 5-35) for the target behavior while responses on the controlled items are summed to form the controlled regulation score (range 8-56). These two subscale scores are used separately.
International Physical Activity Questionnaire Short Version (IPAQ) | June 2018-February 2019.Questionnaires will be completed upon admission to rehabilitation, discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge.
  The IPAQ measures the level of PA across four domains; leisure time PA, domestic and gardening (yard) activities, work- related PA, and transport- related PA. In each domain, the duration (in minutes) and frequency (days) of PA including sitting, walking, moderate and vigorous PA are self-reported.
EuroQol, five dimensions, three levels (EQ-5D-3L) | June 2018-February 2019.Questionnaires will be completed upon admission to rehabilitation, discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge.
  Health related quality of life will be measured using the EuroQol, five dimensions, three levels (EQ-5D-3L). The EQ-5D-3L determines self-assessed problems across five items of mobility, self-care, usual activities, pain/dis- comfort and anxiety/depression. Each item has three levels of severity: 'no problems', 'some problems' and 'severe problems'.
Perceived Competence Scale (Exercising Regularly) | June 2018-February 2019.Questionnaires will be completed upon admission to rehabilitation, discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge.
  The Perceived Competence Scale (PCS) assesses the degree to which patients feel confident about being able to make and maintain their participation in the rehabilitation programme and PA.
Perceived Environmental Supportiveness Scale (PESS) | June 2018-February 2019.Questionnaires will be completed upon admission to rehabilitation, discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge.
  Markland and Tobin (2010) developed the Perceived Environmental Supportiveness Scale (PESS) to assess perceptions of need support provided by exercise practicioners to exercise referral scheme clients. The PESS was designed to explicitly assess the three dimensions of support (autonomy support, structure and involvement) and comprises 15 items with five items assessing each of the three dimensions.
Relatedness to Others in Physical Activity (ROPAS) Scale | June 2018-February 2019.Questionnaires will be completed upon admission to rehabilitation, discharge (on average 8 weeks following admission to rehabilitation), 3 months post-discharge, 6 months post-discharge.
  The Relatedness to Others in Physical Activity Scale (ROPAS) (Wilson & Bengoechea, 2010) will be used to assess participants' perceptions of the group climate. Participants responded to 6-items assessing respondents' perception of meaningful connection and belongingness to other group members. Items are rated on a 6-pt likert scale and a priori criteria for summary scores are set at ≥4.5. An example item includes, "I have developed a close bond with others."
Test of Exercise Capacity | Test will be completed upon admission to rehabilitation, and at discharge (on average 8 weeks following admission to rehabilitation).
  Patients will complete either an Incremental Shuttle Walking Test (ISWT), six-minute walk test (6MWT), or bike test. In all cases, patients' perceived exertion will be assessed with the 15-point single-item Rating of Perceived Exertion (RPE; Borg, 1998), which ranges from 6 (no exertion at all) to 20 (maximal exertion).
Attendance at Rehabilitation Sessions | Throughout rehabilitation programme (on average 8 weeks).
  The number of sessions, over an average of 8 weeks, that each participant attends will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian W Midgley, PhD, Principal Investigator — Liverpool Heart and Chest Hospital NHS Foundation Trust/ Edge Hill University; Bashir Matata, PhD, Principal Investigator — Liverpool Heart and Chest Hospital NHS Foundation Trust
Locations (1):
- Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Arnold E, Bruton A, Ellis-Hill C. Adherence to pulmonary rehabilitation: A qualitative study. Respir Med. 2006 Oct;100(10):1716-23. doi: 10.1016/j.rmed.2006.02.007. Epub 2006 Mar 22. PMID 16554147
- [Background] Bjarnason-Wehrens B, Bott D, Benesch L, Bischoff KO, Buran-Kilian B, Gysan D, Hollenstein U, Mayer-Berger W, Wilkniss R, Sauer G. Long-term results of a three-week intensive cardiac out-patient rehabilitation program in motivated patients with low social status. Clin Res Cardiol. 2007 Feb;96(2):77-85. doi: 10.1007/s00392-007-0461-0. Epub 2006 Dec 14. PMID 17160566
- [Background] British Heart Foundation. (2015). The National Audit of Cardiac Rehabilitation Annual Statistical Report 2015. London. Retrieved from http://www.cardiacrehabilitation.org.uk/docs/2007.pdf
- [Background] British Thoracic Society (BTS). (2013). BTS Guideline on Pulmonary Rehabilitation in Adults. An International Journal of Respiratory Medicine, 68(2), ii1-31. https://doi.org/10.1136/thoraxjnl-2013-203808
- [Background] Chan DK, Lonsdale C, Ho PY, Yung PS, Chan KM. Patient motivation and adherence to postsurgery rehabilitation exercise recommendations: the influence of physiotherapists' autonomy-supportive behaviors. Arch Phys Med Rehabil. 2009 Dec;90(12):1977-82. doi: 10.1016/j.apmr.2009.05.024. PMID 19969157
- [Background] Clark RA, Conway A, Poulsen V, Keech W, Tirimacco R, Tideman P. Alternative models of cardiac rehabilitation: a systematic review. Eur J Prev Cardiol. 2015 Jan;22(1):35-74. doi: 10.1177/2047487313501093. Epub 2013 Aug 13. PMID 23943649
- [Background] De Amici D, Klersy C, Ramajoli F, Brustia L, Politi P. Impact of the Hawthorne effect in a longitudinal clinical study: the case of anesthesia. Control Clin Trials. 2000 Apr;21(2):103-14. doi: 10.1016/s0197-2456(99)00054-9. PMID 10715508
- [Background] Deci, E. L., & Ryan, R. M. (2008). Facilitating optimal motivation and psychological well-being across life's domains. Canadian Psychology/Psychologie Canadienne, 49(1), 14-23. https://doi.org/10.1037/0708-5591.49.1.14
- [Background] Hardcastle SJ, Fortier M, Blake N, Hagger MS. Identifying content-based and relational techniques to change behaviour in motivational interviewing. Health Psychol Rev. 2017 Mar;11(1):1-16. doi: 10.1080/17437199.2016.1190659. Epub 2016 Jun 2. PMID 27189713
- [Background] Hospes G, Bossenbroek L, Ten Hacken NH, van Hengel P, de Greef MH. Enhancement of daily physical activity increases physical fitness of outclinic COPD patients: results of an exercise counseling program. Patient Educ Couns. 2009 May;75(2):274-8. doi: 10.1016/j.pec.2008.10.005. Epub 2008 Nov 25. PMID 19036552
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Moore SM, Charvat JM, Gordon NH, Pashkow F, Ribisl P, Roberts BL, Rocco M. Effects of a CHANGE intervention to increase exercise maintenance following cardiac events. Ann Behav Med. 2006 Feb;31(1):53-62. doi: 10.1207/s15324796abm3101_9. PMID 16472039
- [Background] National Institute for Health and Clinical Excellence (NICE). (2013). Cardiac rehabilitation services: commissioning guide. London.
- [Background] Ntoumanis N, Thogersen-Ntoumani C, Quested E, Hancox J. The effects of training group exercise class instructors to adopt a motivationally adaptive communication style. Scand J Med Sci Sports. 2017 Sep;27(9):1026-1034. doi: 10.1111/sms.12713. Epub 2016 Jun 10. PMID 27283879
- [Background] Prestwich, A., Webb, T. L., & Conner, M. (2015). Using theory to develop and test interventions to promote changes in health behaviour: Evidence, issues, and recommendations. Current Opinion in Psychology, 5(February), 1-5. https://doi.org/10.1016/j.copsyc.2015.02.011
- [Background] Rahman RJ, Thogersen-Ntoumani C, Thatcher J, Doust J. Changes in need satisfaction and motivation orientation as predictors of psychological and behavioural outcomes in exercise referral. Psychol Health. 2011 Nov;26(11):1521-39. doi: 10.1080/08870446.2010.538849. Epub 2011 Jun 16. PMID 22111661
- [Background] Russell KL, Bray SR. Promoting self-determined motivation for exercise in cardiac rehabilitation: the role of autonomy support. Rehabil Psychol. 2010 Feb;55(1):74-80. doi: 10.1037/a0018416. PMID 20175637
- [Background] Silva MN, Vieira PN, Coutinho SR, Minderico CS, Matos MG, Sardinha LB, Teixeira PJ. Using self-determination theory to promote physical activity and weight control: a randomized controlled trial in women. J Behav Med. 2010 Apr;33(2):110-22. doi: 10.1007/s10865-009-9239-y. Epub 2009 Dec 11. PMID 20012179
- [Background] Singh SJ, Smith DL, Hyland ME, Morgan MD. A short outpatient pulmonary rehabilitation programme: immediate and longer-term effects on exercise performance and quality of life. Respir Med. 1998 Sep;92(9):1146-54. doi: 10.1016/s0954-6111(98)90410-3. PMID 9926171
- [Background] Speake H, Copeland RJ, Till SH, Breckon JD, Haake S, Hart O. Embedding Physical Activity in the Heart of the NHS: The Need for a Whole-System Approach. Sports Med. 2016 Jul;46(7):939-46. doi: 10.1007/s40279-016-0488-y. PMID 26942468
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] The Academy of Medical Royal Colleges. (2015). Exercise: The miracle cure and the role of the doctor in promoting it. Report from the Academy of Medical Royal Colleges. London. Retrieved from http://www.aomrc.org.uk
- [Background] Yohannes AM, Doherty P, Bundy C, Yalfani A. The long-term benefits of cardiac rehabilitation on depression, anxiety, physical activity and quality of life. J Clin Nurs. 2010 Oct;19(19-20):2806-13. doi: 10.1111/j.1365-2702.2010.03313.x. Epub 2010 Aug 24. PMID 20738450